CLINICAL TRIAL: NCT00966576
Title: The Efficacy and Safety of Adding the Brinzolamide/Timolol Maleate Fixed Combination (Azarga®) to Prostaglandin Monotherapy
Brief Title: Efficacy and Safety of Adding Azarga to Prostaglandin Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-08-22a
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2012-04

CONDITIONS: Glaucoma
Keywords: Glaucoma; IOP; AZARGA
MeSH Terms: conditions — Glaucoma | interventions — brinzolamide; Azarga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brinzolamide/Timolol Maleate Fixed Combination (Experimental)
  Interventions: Drug: Brinzolamide/Timolol Maleate Fixed Combination (AZARGA)

INTERVENTIONS:
Drug: Brinzolamide/Timolol Maleate Fixed Combination (AZARGA) — 1 drop of study medication into the study eye(s) beginning the evening of Visit 1 and continuing twice daily (morning and evening) for 12 weeks
  Other Names: AZARGA

SUMMARY:
The purpose of this study is to assess the safety and efficacy of adding AZARGA in glaucoma patients with uncontrolled intraocular pressure (IOP), currently on prostaglandin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent.
* 21 years of age or older.
* Able to follow instructions and willing to attend required study visits.
* Clinical diagnosis of ocular hypertension, primary open-angle, or pigment dispersion glaucoma in at least one eye (qualifying eye).
* Intra-ocular pressure (IOP) considered to be safe in both eyes in such a way that should assure clinical stability of vision and the optic nerve throughout the trial.
* Must have best corrected visual acuity of 6/60 (6/60 Snellen, 1.0 LogMAR) or better in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Presence of other primary or secondary glaucomas not listed in inclusion criterion.
* Presence of corneal dystrophies.
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye.
* Intraocular conventional surgery or laser surgery in qualifying eye(s) less than three months prior to Visit 1.
* Risk of visual field or visual acuity worsening as a consequence of participation in the trial, in the investigator's best judgment.
* Women of childbearing potential not using reliable means of birth control.
* Women who are pregnant or lactating.
* Participation in any other investigational study within 30 days prior to Visit 1.
* Current or anticipated use of systemic corticosteroids, by any route except inhaled, for greater than two weeks during the trial.
* Severe allergic rhinitis
* History of ocular herpes simplex.
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The mean decrease in intraocular pressure (IOP) at 12 weeks from baseline | 12 weeks

SECONDARY OUTCOMES:
Safety as determined by visual acuity, biomicroscopy, adverse events, solicited symptom survey and treatment success | Week 4 and Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Mainz, Germany

REFERENCES:
- [Result] Lorenz K, Rosbach K, Matt A, Pfeiffer N. Addition of a fixed combination of brinzolamide 1%/timolol 0.5% to prostaglandin monotherapy in patients with glaucoma or ocular hypertension. Clin Ophthalmol. 2011;5:1745-50. doi: 10.2147/OPTH.S25987. Epub 2011 Dec 9. PMID 22205835